CLINICAL TRIAL: NCT00560274
Title: An Open Label Study to Evaluate the Safety of NeoRecormon in the Treatment of Anemia in Patients With Chronic Hepatitis C Who Are Treated With Pegylated Interferon + Ribavirin Combination Therapy
Brief Title: A Study of NeoRecormon (Epoetin Beta) in Anemic Patients With Chronic Hepatitis C.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21362
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — peginterferon alfa-2a; Ribavirin; epoetin beta

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Pegasys; Drug: Ribavirin; Drug: epoetin beta [NeoRecormon]

INTERVENTIONS:
Drug: Pegasys — As prescribed
Drug: Ribavirin — As prescribed
Drug: epoetin beta [NeoRecormon] — 30,000 IU sc/week (starting dose)

SUMMARY:
This single arm study will assess the safety of NeoRecormon in the correction of anemia in patients with chronic hepatitis C who are being treated with Pegylated interferon + ribavirin combination therapy. Patients will receive NeoRecormon at a starting dose of 30,000 IU s.c. which will be adjusted as required to maintain a target Hb of 11-13g/dL. The anticipated time on study treatment is 1 year, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic hepatitis C;
* quantifiable serum HCV RNA;
* Pegylated interferon + ribavirin treatment started <6 months before study;
* Hb <10g/dL.

Exclusion Criteria:

* treatment with ESA during preceding 12 weeks;
* poorly controlled hypertension;
* history of cancer, except for basal cell cancer and cervical cancer in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2008-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Blood pressure, pulse rate. | 6 and 12 months
AEs, and laboratory parameters. | Throughout study

SECONDARY OUTCOMES:
Percentage of patients achieving correction of anemia | 3 months
Percentage of patients not requiring blood transfusion | 12 months
Course of Hb concentration | 12 months
Percentage of patients maintaining initial ribavirin dose | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- France (21):
  - Angers
  - Besançon
  - Caen
  - Chambray-lès-Tours
  - Clichy
  - Créteil
  - Limoges
  - Lyon
  - Marseille
  - Montpellier
  - Nice
  - Paris
  - Pessac
  - Rennes
  - Rouen
  - Saint-Laurent-du-Var
  - Strasbourg
  - Toulouse
  - Tourcoing
  - Vandœuvre-lès-Nancy
  - Villejuif